CLINICAL TRIAL: NCT05080023
Title: Impact of Enhanced External Counterpulsation (EECP) on Cardiac Force Index
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chi-Ming Chu (Other)
Collaborators: Dr. Chiang, Shang-lin (Unknown); Dr. Liang-Cheng Chen (Unknown)
Responsible Party: Sponsor-Investigator, Chi-Ming Chu, Prof. Dr., National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Other Study IDs: 1-104-05-147
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Enhanced External Counterpulsation (EECP); Cardiac Output; Cardiac Force Index
Keywords: cardiac force index; Cardiac Output; Enhanced External Counterpulsation (EECP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Enhanced External Counterpulsation (EECP) — Enhanced External Counterpulsation (EECP)

SUMMARY:
Regular exercise can prevent cardiovascular disease, but there is also a risk of sudden cardiac death. Exercise-related sudden death often occurs unconsciously and there is no relevant monitoring mechanism. The patent of the Cardiac Force Index (CFI), invented by Professor Chu, is a method to detect the state of cardiac motion. Recent studies have confirmed Enhanced External Counterpulsation (EECP) can increase cardiopulmonary fitness and maximal oxygen consumption. Our aim is to investigate the differences and effects of CFI between two groups with and without 4 weeks of EECP intervention, therefore, to find out the relationship between CFI and maximum oxygen consumption (VO2max).

Methods: A pre and post-test control group was designed. A total of 53 military students (33 males and 20 females) were recruited and divided into intervention and control groups. A 2000-meter running and maximum oxygen consumption tests were performed pre and post-test. The intervention group was conducted a 4 week (3 times per week/30 minutes) EECP intervention.

ELIGIBILITY:
Inclusion Criteria:

* can walk.

Exclusion Criteria:

* disabilities.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects can walk with a cardiac force meter.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Enhanced External Counterpulsation (EECP) on cardiac force index | 4 weeks
  Enhanced External Counterpulsation (EECP) on cardiac force index

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Local Clinics, Hualien City
  - Local Clinics, Kaohsiung City
  - Local Clinics, Taichung
  - National Defense Medical Center, Taipei
  - Local Clinics, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hsiao PJ, Chiu CC, Lin KH, Hu FK, Tsai PJ, Wu CT, Pang YK, Lin Y, Kuo MH, Chen KH, Wu YS, Wu HY, Chang YT, Chang YT, Cheng CS, Chuu CP, Lin FH, Chang CW, Li YK, Chan JS, Chu CM. Usability of Wearable Devices With a Novel Cardiac Force Index for Estimating the Dynamic Cardiac Function: Observational Study. JMIR Mhealth Uhealth. 2020 Jul 21;8(7):e15331. doi: 10.2196/15331. PMID 32706725
- [Background] Chiang KT, Tu MY, Lin YJ, Hsin YH, Chiu YL, Li FL, Chen HH, Lai CY. A Cardiac Force Index Applied to the G Tolerance Test and Surveillance among Male Military Aircrew. Int J Environ Res Public Health. 2021 Aug 21;18(16):8832. doi: 10.3390/ijerph18168832. PMID 34444580